CLINICAL TRIAL: NCT05727033
Title: Extraordinarily Fun Training Project in Compulsory Secondary Education-Sexually Transmitted Infections: Educational Intervention on STI in Adolescents From 1st&2nd Year of Compulsory Secondary Education Incorporating the Gender Perspective
Brief Title: Extraordinarily Fun Training Project in Compulsory Secondary Education - Sexually Transmitted Infections
Acronym: FEDE-ITS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4R22/162
Record Dates: First submitted 2022-11-23; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-11

CONDITIONS: Chlamydia Infections; Gonorrhea; Syphilis Infection; Human Immunodeficiency Virus (HIV); Human Papillomavirus (HPV); Gender Equity
Keywords: Adolescents; sexually transmitted infections; primary health care; sexual health; health education
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Health Education | interventions — Health

STUDY DESIGN:
Intervention Model Description: Cluster randomised clinical trial with the control group, unblinded and with pre-intervention, end-of-intervention and post-intervention assessments six months after the intervention. A 1:1 allocation ratio is established.
Who Masked: Outcomes Assessor
Masking Description: The person in charge of analyzing the data collected in the study will not know if the participants belong to the intervention group or the control group, which will be identified with an alphanumeric code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): The intervention of training-participatory activity will last between 45 and 60 minutes, divided into theoretical training of 15-30 minutes followed by discussion training of 30 minutes. Based on the projection of the posters, photographs and the short film, the pupils will be asked to participate and work on the problem of STIs as well as possible solutions. The group techniques of photo-talk and presentation with a discussion using the short film will be used. Finally, the training includes Kahoot®, a tool for learning and reviewing concepts in a fun, quiz-like way. Four multiple-choice questions have been included. They will learn in a participatory way about STIs, risk practices, barrier methods and health resources to consult or go to in case of suspicion of contracting an STI.
  For the activity, a sequence of drawings and signs has been designed to put STIs, their causes and how to prevent infection into context.
  Interventions: Behavioral: Participatory teaching group
- Control Group (Sham Comparator): Following the indications of the Department of Education and the "Health and School" Programme, non specific training intervention will be carried out in the control group out during the study period.
  Interventions: Behavioral: Sham control group

INTERVENTIONS:
Behavioral: Participatory teaching group — The intervention will be called FEDE-ITS® methodology. This methodology is self-designed and self-developed and draws on previous work in equivalent populations. It is based on teaching in a participatory way knowledge and healthy attitudes related to the five most prevalent STIs in the province of Barcelona and Lleida, the methods to avoid contagion, and the health resources that can be consulted in case of infection, contact with an infected person or concerns. In addition, a gender perspective is incorporated to contribute to freer and more egalitarian relationships and reduce the likelihood of violence against women which develops in adolescence.
  The cross-cutting themes of the training are: health, pleasure, self-esteem, knowledge-based freedom of choice, equality between people and respect for sexual freedom. Therefore, the ultimate goal is to prevent abusive power relations and macho violence.
  Other Names: Extraordinarily Fun Training in compulsory secondary Education - Sexually Transmitted Infections methodology; FEDE-ITS® methodology
  Arms: Intervention Group
Behavioral: Sham control group — The "Health and School" program was implemented to promote health in schools, and for this reason the program's nurse attends annually to address problems related to sexual affective health within the curricular itinerary of each school, but not specifically on sexually transmitted infections or gender perspective.
  Other Names: Sham intervention group; Health and school program (Department of Health. Government of Catalonia)
  Arms: Control Group

SUMMARY:
Project FEDE-ITS will improve the STI knowledge and its treatment, of adolescents in the 1st and 2nd year of compulsory secondary education in the intervention group compared to compared to the control group, and will modify the sexual risk practices and the perception of risky practices of alcohol and other drug use during sex of participants in the intervention group compared to the control group.

DETAILED DESCRIPTION:
Background: Sexually transmitted infections (STIs) are a public health problem. Every day, more than 1 million people are infected worldwide, most of whom are asymptomatic. The most common STIs are chlamydia, gonorrhea, syphilis and trichomoniasis, which are easily curable. Other highly prevalent infections are genital herpes and human papillomavirus. However, there is no clear evidence regarding the effectiveness of interventions. Due to the serious epidemiological situation regarding sexually transmitted infections, actions are needed to mitigate the exponential growth in the incidence of these infections.

Objective: To evaluate the impact of an intervention on sexual education in pupils of 1st and 2nd year of Compulsory Secondary Education (ESO), assessing the knowledge about the five most prevalent STIs, the knowledge of barrier methods, and practice of STI risky behaviours.In addition, to analyze whether biological sex conditions the role of submission in women versus the role of dominance in men.

Trial Design: Cluster randomised clinical trial.

Location: It will be carried out in the Basic Health Area of Sant Andreu de la Barca (Baix Llobregat Nord), Balaguer (Noguera), Alcarràs (Segrià) and Barcelona (Barcelona), in Catalonia, Spain.

Participants: Students enrolled in secondary education schools in ESO 1st and 2nd years who meet the selection criteria.

Instruments: As an intervention to be evaluated, an innovative educational methodology with a gender perspective will be carried out on adolescents through discussion with photographs, posters and a short film. No training intervention will be carried out in the control group during the study period, following the instructions of the Department of Education of the Generalitat of Catalonia.

Variables: Evaluation in both groups of knowledge, attitudes and risk practices related to STIs through a pre-intervention, post-intervention and post-post-intervention questionnaire validated in previous studies.

Applicability: The aim is to explore new educational methods to improve knowledge, attitudes and risk practices for STIs in future sexual relationships. Gender-sensitive training could contribute to freer and more egalitarian relationships and reduce the likelihood of violence against women that develops in adolescence.

ELIGIBILITY:
Inclusion Criteria:

* pupils in the 1st and 2nd years of compulsory secondary education in the municipalities of Sant Andreu de la Barca, Balaguer, Alcarràs and Barcelona
* prior authorisation of the school administration,
* prior authorisation of the pupil
* prior authorisation of the parents/legal guardians by submitting the information sheet and collecting the informed consent.

Exclusion Criteria:

* pupils refusing to participate
* families refusing to participate
* school administration refusing to participate

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Knowledge of the five most prevalent STIs | pre-intervention at the baseline day
  Discrete quantitative variable. It will be assessed by scoring. 5 scoring items: correct answer 1 point and incorrect answer 0 points. The maximum score will be 5 points (HIV: 1 point, Chlamydia: 1 point, Syphilis or Treponema pallidum: 1 point, Gonorrhoea or Neisseria gonorrhoeae: 1 point, HPV or Papilloma Virus: 1 point), and the minimum 0 points.
  - "List the Sexually Transmitted Infections (STIs) you know, Tick one:
  * HIV
  * Candida albicans
  * Gonorrhoea
  * Chlamydia
  * Escherichia coli
  * Treponema / Syphilis
  * COVID-19
  * Human Papilloma (HPV)"
Knowledge of the five most prevalent STIs | end-of-intervention at the same day
  Discrete quantitative variable. It will be assessed by scoring. 5 scoring items: correct answer 1 point and incorrect answer 0 points. The maximum score will be 5 points (HIV: 1 point, Chlamydia: 1 point, Syphilis or Treponema pallidum: 1 point, Gonorrhoea or Neisseria gonorrhoeae: 1 point, HPV or Papilloma Virus: 1 point), and the minimum 0 points.
  - "List the Sexually Transmitted Infections (STIs) you know, Tick one:
  * HIV
  * Candida albicans
  * Gonorrhoea
  * Chlamydia
  * Escherichia coli
  * Treponema / Syphilis
  * COVID-19
  * Human Papilloma (HPV)"
Knowledge of the five most prevalent STIs | post-intervention assessments six months after the intervention
  Discrete quantitative variable. It will be assessed by scoring. 5 scoring items: correct answer 1 point and incorrect answer 0 points. The maximum score will be 5 points (HIV: 1 point, Chlamydia: 1 point, Syphilis or Treponema pallidum: 1 point, Gonorrhoea or Neisseria gonorrhoeae: 1 point, HPV or Papilloma Virus: 1 point), and the minimum 0 points.
  - "List the Sexually Transmitted Infections (STIs) you know, Tick one:
  * HIV
  * Candida albicans
  * Gonorrhoea
  * Chlamydia
  * Escherichia coli
  * Treponema / Syphilis
  * COVID-19
  * Human Papilloma (HPV)"
Knowledge of different barrier methods. | pre-intervention at the baseline day
  Discrete quantitative variable. It will be collected in the questionnaire using a question with multiple correct options. There will be 5 options and 2 correct. Scoring: From 0 (minimum score) to 5 points (maximum score)
  - "How many barrier methods do you know? (tick the options you consider * correct): Select all the options that apply.
  * Male condom
  * Post-coital pill
  * Aspirin
  * Abstinence
  * Female condom"
Knowledge of different barrier methods. | end-of-intervention at the same day
  Discrete quantitative variable. It will be collected in the questionnaire using a question with multiple correct options. There will be 5 options and 2 correct. Scoring: From 0 (minimum score) to 5 points (maximum score)
  - "How many barrier methods do you know? (tick the options you consider * correct): Select all the options that apply.
  * Male condom
  * Post-coital pill
  * Aspirin
  * Abstinence
  * Female condom"
Knowledge of different barrier methods. | post-intervention assessments six months after the intervention
  Discrete quantitative variable. It will be collected in the questionnaire using a question with multiple correct options. There will be 5 options and 2 correct. Scoring: From 0 (minimum score) to 5 points (maximum score)
  - "How many barrier methods do you know? (tick the options you consider * correct): Select all the options that apply.
  * Male condom
  * Post-coital pill
  * Aspirin
  * Abstinence
  * Female condom"
Use of barrier methods in sexual intercourse. | pre-intervention at the baseline day
  Ordinal qualitative variable. It will be recorded in the questionnaire using a Likert scale (always, almost always, sometimes, never)
  - In the case of having sex, have you used barrier methods (condom or female condom) from the very start (including oral sex), OR If you do not have sex, do you think that when you do have sex you will always use barrier methods (condom-female condom), including oral sex? Tick one.
  * Always
  * Almost Always
  * Sometimes
  * Never
Use of barrier methods in sexual intercourse. | end-of-intervention at the same day
  Ordinal qualitative variable. It will be recorded in the questionnaire using a Likert scale (always, almost always, sometimes, never)
  - In the case of having sex, have you used barrier methods (condom or female condom) from the very start (including oral sex), OR If you do not have sex, do you think that when you do have sex you will always use barrier methods (condom-female condom), including oral sex? Tick one.
  * Always
  * Almost Always
  * Sometimes
  * Never
Use of barrier methods in sexual intercourse. | post-intervention assessments six months after the intervention
  Ordinal qualitative variable. It will be recorded in the questionnaire using a Likert scale (always, almost always, sometimes, never)
  - In the case of having sex, have you used barrier methods (condom or female condom) from the very start (including oral sex), OR If you do not have sex, do you think that when you do have sex you will always use barrier methods (condom-female condom), including oral sex? Tick one.
  * Always
  * Almost Always
  * Sometimes
  * Never
Drug use during sexual intercourse. | pre-intervention at the baseline day
  Qualitative ordinal variable. It will be recorded in the questionnaire using a Likert scale (always, almost always, sometimes, never)
  - "If you have sex, do you use alcohol or other drugs when you have sex? OR If you do not have sex, do you think that when you do you will use * alcohol or other drugs when you have sex? Tick one.
  * Always
  * Almost Always
  * Sometimes
  * Never
Drug use during sexual intercourse. | end-of-intervention at the same day
  Qualitative ordinal variable. It will be recorded in the questionnaire using a Likert scale (always, almost always, sometimes, never)
  - "If you have sex, do you use alcohol or other drugs when you have sex? OR If you do not have sex, do you think that when you do you will use * alcohol or other drugs when you have sex? Tick one.
  * Always
  * Almost Always
  * Sometimes
  * Never
Drug use during sexual intercourse. | post-intervention assessments six months after the intervention
  Qualitative ordinal variable. It will be recorded in the questionnaire using a Likert scale (always, almost always, sometimes, never)
  - "If you have sex, do you use alcohol or other drugs when you have sex? OR If you do not have sex, do you think that when you do you will use * alcohol or other drugs when you have sex? Tick one.
  * Always
  * Almost Always
  * Sometimes
  * Never

SECONDARY OUTCOMES:
Role in sexual intercourse. | pre-intervention at the baseline day
  Nominal qualitative variable. It will be recorded in the questionnaire using multiple-choice questions.
  "If you have sex, who decides whether or not to use a barrier method of contraception (condom - female condom)? OR If you do not have sex, who do you think will decide whether or not to use * a barrier method of contraception (condom-female condom) when you do have sex Tick one.
  * Myself
  * My sexual partner
  * We decide by mutual consent
  * Other (specify)
Role in sexual intercourse. | end-of-intervention at the same day
  Nominal qualitative variable. It will be recorded in the questionnaire using multiple-choice questions.
  "If you have sex, who decides whether or not to use a barrier method of contraception (condom - female condom)? OR If you do not have sex, who do you think will decide whether or not to use * a barrier method of contraception (condom-female condom) when you do have sex Tick one.
  * Myself
  * My sexual partner
  * We decide by mutual consent
  * Other (specify)
Role in sexual intercourse. | post-intervention assessments six months after the intervention
  Nominal qualitative variable. It will be recorded in the questionnaire using multiple-choice questions.
  "If you have sex, who decides whether or not to use a barrier method of contraception (condom - female condom)? OR If you do not have sex, who do you think will decide whether or not to use * a barrier method of contraception (condom-female condom) when you do have sex Tick one.
  * Myself
  * My sexual partner
  * We decide by mutual consent
  * Other (specify)

CONTACTS AND LOCATIONS:
Overall Officials: David Pedrazas-López, PhD, MD, Principal Investigator — Institut Català de la Salut
Locations (4):
- Spain (4):
  - CAP Sant Andreu de la Barca, Sant Andreu de la Barca, Barcelona
  - CAP Alcarràs, Alcarràs, Lleida
  - CAP Balaguer, Balaguer, Lleida
  - CAP Gótic, Barcelona

IPD SHARING:
Plan to Share IPD: No